CLINICAL TRIAL: NCT01327196
Title: Detection of Mild Cognitive Impairment in People Older Than 65 Years of Age and Its Relationship to Cardiovascular Risk Factors (DECRIVAM)
Brief Title: Cognitive Impairment and Cardiovascular Risk in Older
Acronym: DECRIVAM
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Grupo de Investigación de Atención Primaria de Castilla y León (Other Government)
Responsible Party: Sponsor
Other Study IDs: BIO39/SA04/10
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2014-09

CONDITIONS: Cognitive Impairment; Cardiovascular Risk Factor
Keywords: dementia; cardiovascular risk; elderly; aging; older 65-100 years
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this project is to study cognitive yields in people of the town of Salamanca over 65, with particular emphasis on the acquisition of the initial symptoms of cognitive impairment in order to detect mild cognitive impairment and study the relationship between the clinical situation and cardiovascular risk factors. It will depart from a reference population of 420 people older than 65 years living in the municipality of Salamanca which took part in a survey prior to partner health needs of the elderly of 65 years in the municipality of Salamanca. This was a stratified sampling as stratum considering the area of health. The results of this study are expected to evidence the extent of the problem of cognitive decline in the population over 65 years. It is also expected to determine the relationship between the co-morbidity in this problem and specific factors of cardiovascular risk in this group of population.

DETAILED DESCRIPTION:
A random sample population, the information obtained has a validity superior to other studies in which the sample has not followed very strict criteria of selection.

Protocol for measurement:

* variable demographic partner
* vascular risk factors
* co-morbidity
* functional level for the activities of daily life
* cognitive performance in attention, memory, language, praxias, gnosias (abbreviated neuropsychological battery)

Through a battery short neuropsychological specially adapted for the study of older people will carry out a study of the cognitive performance in people older than 65 years of age and will try to establish how much influence the controlled variables of cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* lives in the municipality of Salamanca
* over 65 years of age

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: It will depart from a reference population of 420 people older than 65 years living in the municipality of Salamanca
Sampling Method: Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of risk factors cardiovascular | Prevalence of risk factors cardiovascular

SECONDARY OUTCOMES:
neuropsychological assessment | neuropsychological assessment

OTHER OUTCOMES:
neuropsychological assessment | neuropsychological assessment

CONTACTS AND LOCATIONS:
Overall Officials: MºVictoria Perea-Bartolome, MD, Principal Investigator — Fundacion INFOSALUD; Emiliano Rodriguez-Sanchez, MD, Study Director — Fundacion INFOSALUD
Locations (1):
- Fundacion INFOSALUD, Salamanca, Spain

REFERENCES:
- [Derived] Perea-Bartolome MV, Garcia-Garcia R, Ladera-Fernandez V, Mora-Simon S, Patino-Alonso MC, Almanza-Guerra TJ, Agudo-Conde C, Muriel-Diez MP, Rodriguez-Sanchez E. Detection of mild cognitive impairment in people older than 65 years of age and its relationship to cardiovascular risk factors (DECRIVAM). BMC Public Health. 2011 Jun 27;11:504. doi: 10.1186/1471-2458-11-504. PMID 21708036